CLINICAL TRIAL: NCT04319679
Title: The Effects of Extracorporeal Shockwave Therapy (ESWT) for Upper Extremity Pain Related to Spasticity in Patients With Spinal Cord Injury
Brief Title: ESWT for UE Pain in Patients With Cervical Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, MinYoung Kim, MD, PhD, Principal Professor of Rehabilitation Medicine, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESWTSCIPain
Record Dates: First submitted 2020-03-14; First posted 2020-03-24 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Spastic Tetraplegia; Pain; Myelopathy Cervical
Keywords: Extracorporeal shockwave therapy; Cervical myelopathy; Spasticity; Pain
MeSH Terms: conditions — Quadriplegia; Pain; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 3,000 pulses per time, low energy under 0.3 mJ/mm^2, tolerable range
  Interventions: Device: Extracorporeal shockwave therapy
- Control group (Sham Comparator): Sham therapy
  Interventions: Device: Sham therapy

INTERVENTIONS:
Device: Extracorporeal shockwave therapy — 6 times during 2 weeks
  Arms: Experimental group
Device: Sham therapy — 6 times during 2 weeks
  Arms: Control group

SUMMARY:
This study aimed to investigate the efficacy and safety of extracorporeal shockwave therapy (ESWT) for upper extremity pain related to spasticity in patients with spinal cord injury.

DETAILED DESCRIPTION:
6 times of ESWT (3,000 pulses per time, low energy under 0.3 mJ/m^2, tolerable range) on forearm area to reduce pain related to spasticity in patients with cervical myelopathy

ELIGIBILITY:
Inclusion Criteria:

1. Spinal cord damage confirmed in the spinal cord image
2. 1 month after spinal cord injury
3. Spasticity of upper extremities
4. Pain in areas below spinal cord injury more than 4 points on the numerical scale (NRS)
5. Cognitive functions that can clearly point out NRS with more than 15 points in the mini mental state examination (MMSE)
6. Age: 20 and older
7. Person who has agreed in writing to decide his or her participation and comply with the precautions

Exclusion Criteria:

1. Pain due to trauma
2. Injection treatments two weeks before participating in the study
3. Severe coagulopathy (excluding antiplatelet use)
4. Impaired cognition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | Up to 4 weeks (baseline, after each treatment during 2 weeks, 2 weeks + 1 day, 4 weeks)
  Pain intensity (0-10, ordinal scale)

SECONDARY OUTCOMES:
Modified Ashworth scale (MAS) | Up to 4 weeks (baseline, after each treatment during 2 weeks, 2 weeks + 1 day, 4 weeks)
  Spasticity, ordinal scale (0, 1, 1+, 2, 3, 4: higher scores indicate more severe spasticity)
Range of motion (ROM) | Up to 4 weeks (baseline, 1 week, 2 weeks, 2 weeks + 1 day, 4 weeks)
  Passive ROM of elbow, wrist and 3rd finger (in degrees: higher scores indicate larger range)
Grasp power | Up to 4 weeks (baseline, 2 weeks, 4 weeks)
  Hand grip power (in Kg measured by a dynamometer: higher scores indicate stronger power)

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghoon Min, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, CHA Bundang Medical Center, CHA University School of Medicine
Locations (1):
- Department of Rehabilitation Medicine, CHA Bundang Medical Center,, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Information that cannot be identified
Supporting Information: Study Protocol